CLINICAL TRIAL: NCT00524368
Title: A Randomized, Open-label Trial to Compare the Efficacy, Safety and Tolerability of DRV/Rtv (800mg/100mg) q.d Versus DRV/Rtv (600mg/100mg) b.i.d in Early Treatment-experienced HIV-1 Infected Subjects
Brief Title: A Study to Compare Effectiveness and Safety of Darunavir/Ritonavir (DRV/Rtv) 800mg/100mg Once Daily Versus DRV/Rtv 600mg/100mg Twice Daily in Early Treatment-Experienced HIV-1 Infected Patients (ODIN)
Acronym: ODIN
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Tibotec Pharmaceuticals, Ireland (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR013783; TMC114-TiDP31-C229 (Other: Tibotec Pharmaceuticals, Ireland); 2007-001939-61 (EudraCT Number); NCT00613990 (obsolete NCT alias)
Record Dates: First submitted 2007-08-30; First posted 2007-09-03 (Estimated); Results first posted 2010-09-22 (Estimated); Last update posted 2013-02-15 (Estimated); Status verified 2013-02

CONDITIONS: Human Immunodeficiency Virus - Type 1
Keywords: Human immunodeficiency virus - type 1; HIV-1 Infection; TMC-114; Darunavir; Ritonavir
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome | interventions — Darunavir; Ritonavir

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- DRV/rtv 800/100 mg once daily (Experimental): Two 400 mg darunavir (DRV) ie, TMC114 tablets + one 100 mg ritonavir (rtv) capsule once daily.
  Interventions: Drug: Darunavir (DRV); Drug: Ritonavir (rtv)
- DRV/rtv 600/100 mg twice daily (Experimental): One 600 mg TMC114 tablet + one 100 mg capsule of rtv twice daily.
  Interventions: Drug: Darunavir (DRV); Drug: Ritonavir (rtv)

INTERVENTIONS:
Drug: Darunavir (DRV) — DRV/rtv 800/100 mg once daily group: 2 tablets of 400 mg of DRV administered orally once daily. DRV/rtv 600/100 mg twice daily group: 1 tablet of 600 mg DRV administered orally twice daily.
  Other Names: TMC114
Drug: Ritonavir (rtv) — DRV/rtv 800/100 mg once daily group: One capsule of 100 mg of ritonavir administered orally once daily. DRV/rtv 600/100 mg twice daily group: One capsule of 100 mg of ritonavir administered orally twice daily.
  Other Names: rtv

SUMMARY:
The purpose of this study is to test if being treated with darunavir/ritonavir (DRV/rtv) 800/100 mg daily is as effective as being treated with DRV/rtv 600/100 mg twice daily, in early antiretroviral (ARV)-experienced patients when given along with selected optimized background regimen (OBR).

DETAILED DESCRIPTION:
This is a randomized (the study medication is assigned by chance), open-label (all people know the identity of the intervention) study in which 590 patients will be randomly assigned to receive either DRV/rtv 800/100 mg daily or DRV/rtv 600/100 mg twice daily along with the selected OBR. An OBR will consist of at least 2 nucleoside reverse transcriptase inhibitors (NRTIs) selected by the investigator. The study will include a 4 week screening period, 48-weeks of treatment period and 4-weeks of follow-up. The study will also consists of extension phase after Week 48: in regions where DRV is not yet commercially available or reimbursed by the health care system, patients who complete the 48 weeks of treatment with DRV/rtv and who continue to benefit from this treatment, will have the opportunity to continue DRV treatment as a 600 mg twice daily dosage until DRV is reimbursed and available via the public and/or private health care system or until its development is discontinued. Safety evaluation will consists of adverse events (including specific toxicities), clinical laboratory tests, vital signs, electrocardiogram, physical and skin examination.

ELIGIBILITY:
Inclusion Criteria:

* Patients with documented human immunodeficiency virus - Type 1 (HIV-1) infection
* Patients with a viral load greater than 1,000 HIV-1 ribonucleic acid (RNA) copies/mL
* Stable highly active antiretroviral therapy (HAART) regimen for at least 12 weeks at screening
* In the investigator's opinion, non-nucleoside reverse transcriptase inhibitors (NNRTIs) are not a valid treatment option, because of the patient's antiretroviral (ARV) treatment history, ARV resistance testing, medication-taking behavior, safety and tolerability concerns, or other patient-related factors
* Prescreening or/and screening plasma HIV-1 RNA greater than 1,000 copies/mL on HAART regimen at screening

Exclusion Criteria:

* Presence of any currently active conditions that fit the definition of the World Health Organization (WHO) Clinical Stage 4, with the following exceptions: stable cutaneous kaposi's sarcoma (ie, no internal organ involvement other than oral lesions) that is unlikely to require any form of systemic therapy during the study time period, wasting syndrome
* Patients for whom an investigational ARV is part of the current regimen, with the following exceptions if applicable (depending on local regulatory approval): tenofovir, emtricitabine
* Previous or current use of enfuvirtide (ENF), tipranavir and/or DRV
* Life expectancy of less than 12 months
* Pregnant or breast-feeding females
* Any active clinically significant disease (eg, tuberculosis [TB], cardiac dysfunction, pancreatitis, acute viral infections) or findings during screening of medical history or physical examination that, in the investigator's opinion, would compromise the patient's safety or outcome of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 590 (Actual)
Dates: Start 2007-10; Primary Completion 2009-08 (Actual); Study Completion 2011-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tibotec Pharmaceuticals, Ireland Clinical Trial, Study Director — Tibotec Pharmaceuticals, Ireland
Locations (85):
- United States (30):
  - Phoenix, Arizona
  - Little Rock, Arkansas
  - Beverly Hills, California
  - Oakland, California
  - Palm Springs, California
  - Fort Lauderdale, Florida
  - Fort Laudersale, Florida
  - Miami, Florida
  - Miami Beach, Florida
  - Orlando, Florida
  - Safety Harbor, Florida
  - West Palm Beach, Florida
  - Atlanta, Georgia
  - Macon, Georgia
  - Savannah, Georgia
  - Chicago, Illinois
  - Springfield, Massachusetts
  - Berkley, Michigan
  - Newark, New Jersey
  - Albany, New York
  - New York, New York
  - Rochester, New York
  - The Bronx, New York
  - Huntersville, North Carolina
  - Winston-Salem, North Carolina
  - Akron, Ohio
  - Charleston, South Carolina
  - Dallas, Texas
  - Harlingen, Texas
  - Houston, Texas
- Argentina (5):
  - Buenos Aires
  - Córdoba
  - Guernica
  - Neuquén
  - Rosario
- Australia (2):
  - Darlinghurst
  - Surry Hills
- Vienna, Austria
- Brazil (7):
  - Curitiba
  - Distrito Barao Geraldo-Campina
  - Pinheiros
  - Recife
  - Rio de Janeiro
  - Salvador
  - São Paulo
- Chile (2):
  - Providencia
  - Santiago
- France (5):
  - Lyon
  - Nice
  - Orléans
  - Paris
  - Vandœuvre-lès-Nancy
- Germany (3):
  - Berlin
  - Cologne
  - München
- Guatemala City, Guatemala
- Budapest, Hungary
- Malaysia (4):
  - Ipoh
  - Kuala Lumpur
  - Pulau Pinang
  - Sungai Buloh
- Panama City, Panama
- San Juan, Puerto Rico
- Romania (4):
  - Bucharest
  - Constanța
  - Iași
  - Timișoara
- South Africa (8):
  - Cape Town
  - Cyrildene Johannesburg Gauteng
  - Dundee
  - Durban
  - Houghton, Johannesburg
  - Johannesburg
  - Pretoria
  - Westdene Johannesburg Gauteng
- Spain (2):
  - Barcelona
  - Madrid
- Taiwan (3):
  - Kaohsiung County
  - Taichung
  - Taipei
- Thailand (4):
  - Bangkok
  - Chiang Mai
  - Khon Kaen
  - Nonthaburi
- London, United Kingdom

REFERENCES:
- [Derived] Lathouwers E, De La Rosa G, Van de Casteele T, Baeten B, Tomaka F, De Meyer S, Picchio G. Virological analysis of once-daily and twice-daily darunavir/ritonavir in the ODIN trial of treatment-experienced patients. Antivir Ther. 2013;18(3):289-300. doi: 10.3851/IMP2569. Epub 2013 Apr 4. PMID 23558157

RESULTS

PARTICIPANT FLOW:
Recruitment Details: One hundred thirteen investigators in 21 countries participated in this study.
Pre-assignment Details: In total 1092 participants were screened, of which 590 participants were randomly assigned and treated (294 participants were treated with DRV/rtv 800/100 mg once daily, and 296 participants with DRV/rtv 600/100 mg twice daily.
Groups:
- DRV/Rtv 800/100 mg Once Daily: Two 400 mg tablets of darunavir (DRV) + one 100 mg capsule of ritonavir (rtv) once daily
- DRV/Rtv 600/100 mg Twice Daily: One 600 mg darunavir (DRV) tablet + one 100 mg capsule of ritonavir (rtv) given twice daily
Period: Overall Study
Arm/Group | DRV/Rtv 800/100 mg Once Daily | DRV/Rtv 600/100 mg Twice Daily
Started | 294 | 296
Completed | 253 | 248
Not Completed | 41 | 48
Not completed — Adverse Event | 10 | 12
Not completed — Lost to Follow-up | 9 | 13
Not completed — Withdrawal by Subject | 4 | 5
Not completed — Non-compliant | 8 | 9
Not completed — Reached a Virologic Endpoint | 3 | 2
Not completed — Sponsor's Decision | 2 | 0
Not completed — Ineligible to Continue the study | 2 | 5
Not completed — Other | 3 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | DRV/Rtv 800/100 mg Once Daily | DRV/Rtv 600/100 mg Twice Daily | Total
Number analyzed (Participants) | 294 | 296 | 590
Age Continuous [Mean (Standard Deviation); unit: years] | 40.2 (9.09) | 40.7 (9.50) | 40.5 (9.29)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 115 | 98 | 213
  Male | 179 | 198 | 377
Age (years) (categorical) [Number; unit: participants]
  Age <= 30 | 35 | 35 | 70
  30 < Age <= 45 | 180 | 169 | 349
  45 < Age <= 55 | 64 | 72 | 136
  55 < Age <= 65 | 14 | 18 | 32
  Age > 65 | 1 | 2 | 3
Hepatitis B or C Co-infection Status [Number; unit: participants]
  Negative | 267 | 255 | 522
  Positive | 25 | 37 | 62
  Unknown | 2 | 4 | 6

OUTCOME MEASURES:

1. Primary Outcome: Virological Response at Week 48 (Number of Participants With Plasma Viral Load Less Than 50 Copies/mL) - as Defined by the Time to Loss of Virologic Response (TLOVR) Algorithm
Description: The TLOVR algorithm was used to derive response, ie, response and loss of response needed to be confirmed at 2 consecutive visits and participants who permanently discontinued were considered nonresponders after discontinuation. Participants with intermittent missing viral load values were considered responders if the preceeding and succeeding visits indicated response. In all other cases, intermittent values were imputed with nonresponse. Resuppression after confirmed virologic failure was considered as failure in this algorithm.
Time Frame: 48 Weeks
Population: Intention To Treat (ITT) population: Participants who permanently discontinued were considered nonresponders after discontinuation. Participants with intermittent missing viral load values were considered responders if preceeding and succeeding visits indicated response. Otherwise, intermittent values were imputed with nonresponse.
Measure: Number; unit: Participants
Arm/Group | DRV/Rtv 800/100 mg Once Daily | DRV/Rtv 600/100 mg Twice Daily
Number analyzed (Participants) | 294 | 296
Participants | 212 | 210
Statistical Analysis 1: Comparison: DRV/Rtv 800/100 mg Once Daily vs DRV/Rtv 600/100 mg Twice Daily; Assuming a response rate of 70% at 48 weeks for both treatment groups, 306 participants were required per treatment arm to establish noninferiority of darunavir (DRV)/ritonavir (rtv) once daily versus DRV/rtv twice daily with a maximum allowable difference of 12%, with a 1-sided significance level of 0.025 and 90% power; Test type: Non-Inferiority or Equivalence — If at Week 48, the lower limit of the 95% two-sided confidence interval of the difference between DRV/rtv once daily and DRV/rtv twice daily exceeds -12%, non-inferiority of the DRV/rtv q.d. versus the DRV/rtv b.i.d. therapy was concluded; p < 0.001, Regression, Logistic; The model includes treatment as factor and baseline viral load (log10) as covariate; Difference in proportion of response = 0.0019, 95% CI 2-sided [-0.054 to 0.092], Standard Error of Mean 0.037 — Difference in proportion of response DRV/rtv once daily minus DRV/rtv twice daily estimated from the logistic regression model

2. Secondary Outcome: Virologic Response at Week 48 (Viral Load Less Than 400 Copies/mL)
Description: Number of participants with confirmed plasma viral load less than 400 copies/mL at Week 48.
Time Frame: 48 weeks
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | DRV/Rtv 800/100 mg Once Daily | DRV/Rtv 600/100 mg Twice Daily
Number analyzed (Participants) | 294 | 296
Participants | 226 | 227
Statistical Analysis 1: Comparison: DRV/Rtv 800/100 mg Once Daily vs DRV/Rtv 600/100 mg Twice Daily; Test type: Non-Inferiority or Equivalence — If at Week 48, the lower limit of this 95% 2-sided CI of the difference between DRV/rtv q.d. and DRV/rtv b.i.d. exceeded -12%, noninferiority of DRV/rtv q.d. and DRV/rtv b.i.d. could be concluded; p < 0.001, Regression, Logistic; A logistic regression model includes treatment as fixed factor and baseline plasma viral load as a covariate; Difference in proportion of response = 0.007, 95% CI 2-sided [-0.060 to 0.075], Standard Error of Mean 0.034 — Difference in proportion of response between 2 treatment groups (DRV/rtv q.d. minus DRV/rtv b.i.d)

3. Secondary Outcome: Change in log10 Viral Load From Baseline at Week 48
Time Frame: 48 weeks
Population: as for outcome 1
Measure: Median (Full Range); unit: log10 copies/mL
Arm/Group | DRV/Rtv 800/100 mg Once Daily | DRV/Rtv 600/100 mg Twice Daily
Number analyzed (Participants) | 294 | 296
log10 copies/mL
  Log10 Viral Load at baseline | 4.23 [1.73 to 6.43] | 4.134 [1.69 to 5.98]
  Log10 Viral Load change from baseline at Week 48 | -2.11 [-4.7 to 2.0] | -2.13 [-4.2 to 2.4]
Statistical Analysis 1: Comparison: DRV/Rtv 800/100 mg Once Daily vs DRV/Rtv 600/100 mg Twice Daily; Test type: Superiority or Other; p = 0.977, ANCOVA; Including 1 factor for treatment, and including the covariate baseline log10 plasma viral load; Difference between least square means = -0.003, 95% CI 2-sided [-0.188 to 0.182], Standard Error of Mean 0.094 — Difference between least square means between the DRV/rtv q.d. and DRV/rtv b.i.d. treatment groups at Week 48

4. Secondary Outcome: Time to Reach First Virologic Response
Description: Time (in weeks) to achieve viral load less than 50 copies/mL by the participants.
Time Frame: 48 weeks
Population: as for outcome 1
Measure: Median (Full Range); unit: Days
Arm/Group | DRV/Rtv 800/100 mg Once Daily | DRV/Rtv 600/100 mg Twice Daily
Number analyzed (Participants) | 294 | 296
Days | 85 [71 to 86] | 85 [83 to 85]
Statistical Analysis 1: Comparison: DRV/Rtv 800/100 mg Once Daily vs DRV/Rtv 600/100 mg Twice Daily; Test type: Superiority or Other; p = 0.917, Cox proportional hazards; Including treatment as fixed factor and baseline plasma viral load as a covariate; Hazard Ratio (HR) = 0.990, 95% CI 2-sided [0.824 to 1.191], Standard Error of Mean 0.094

5. Secondary Outcome: Time to Loss of Virologic Response
Description: Time taken to lose the virologic response ie, plasma viral load less than 50 copies/mL by participants.
Time Frame: 48 weeks
Population: as for outcome 1
Measure: Mean (Standard Error); unit: Days
Arm/Group | DRV/Rtv 800/100 mg Once Daily | DRV/Rtv 600/100 mg Twice Daily
Number analyzed (Participants) | 294 | 296
Days | 250.235 (6.598) | 281.743 (7.47)
Statistical Analysis 1: Comparison: DRV/Rtv 800/100 mg Once Daily vs DRV/Rtv 600/100 mg Twice Daily; Test type: Superiority or Other; p = 0.716, Regression, Cox; Including baseline log10 viral load as covariate; Hazard Ratio, log = 0.945, 95% CI 2-sided [0.699 to 1.279], Standard Error of Mean 0.154

6. Secondary Outcome: Time-averaged Difference (DAVG) of log10 Plasma Viral Load Over 48 Weeks
Time Frame: 48 weeks
Population: Intention To Treat (ITT) population: Observed cases
Measure: Least Squares Mean (Standard Error); unit: log10 copies/mL
Arm/Group | DRV/Rtv 800/100 mg Once Daily | DRV/Rtv 600/100 mg Twice Daily
Number analyzed (Participants) | 294 | 296
log10 copies/mL | -1.77 (0.051) | -1.74 (0.051)
Statistical Analysis 1: Comparison: DRV/Rtv 800/100 mg Once Daily vs DRV/Rtv 600/100 mg Twice Daily; Test type: Superiority or Other; p = 0.711, ANCOVA; Including 1 factor for treatment, and including the covariate baseline log10 plasma viral load; Difference in least square means = -0.03, 95% CI 2-sided [-0.169 to 0.115], Standard Error of Mean 0.072 — Difference in least square means between the 2 treatment groups (DRV/rtv q.d. and DRV/rtv b.i.d)

7. Secondary Outcome: Change in CD4+ Cell Count From Baseline
Description: CD4+ cell count was calculated using the Last Observation Carried Forward (LOCF) algorithm.
Time Frame: 48 Weeks
Population: Intention To Treat (ITT) population - last observation carried forward (LOCF): Intermittent missing values and missing values due to premature discontinuation were imputed with the last observation.
Measure: Median (Full Range); unit: 10e6/l
Arm/Group | DRV/Rtv 800/100 mg Once Daily | DRV/Rtv 600/100 mg Twice Daily
Number analyzed (Participants) | 294 | 296
10e6/l
  Value at Baseline | 219 [24 to 1306] | 236 [44 to 864]
  CD4+ cell count change from baseline at Week 48 | 100 [-242 to 808] | 94 [-239 to 639]
Statistical Analysis 1: Comparison: DRV/Rtv 800/100 mg Once Daily vs DRV/Rtv 600/100 mg Twice Daily; Test type: Superiority or Other; p = 0.562, ANCOVA; The model includes treatment as factor and baseline CD4 count and baseline viral load (log10) as covariates; Difference in least square means = -5.95, 95% CI 2-sided [-26.09 to 14.20], Standard Error of Mean 10.26 — Difference in least square means DRV/rtv once daily minus DRV/rtv twice daily estimated from the ANCOVA model

8. Secondary Outcome: Change From Baseline in Total Functional Assessment of HIV Infection (FAHI) Score
Description: The FAHI is a 44-item questionnaire and incorporates 5 functional scales (physical well-being, emotional well-being/living with HIV, functional and global well-being, social well-being, and cognitive functioning). Each scale included several questions (all 5 scales include total 44 questions). For each question, participants gave a score of either 0 (not at all), 1 (a little bit), 2 (somewhat), 3 (quite a bit) and 4 (very much). Total FAHI imputed score is calculated by adding scores for each question. The range of total FAHI score is 0 to 176. Higher scores indicate worsening.
Time Frame: 48 weeks
Population: as for outcome 7
Measure: Median (Full Range); unit: Scores on a scale
Arm/Group | DRV/Rtv 800/100 mg Once Daily | DRV/Rtv 600/100 mg Twice Daily
Number analyzed (Participants) | 294 | 296
Scores on a scale
  FAHI score at baseline | 129 [31 to 175] | 123.5 [33 to 174]
  Change from baseline in FAHI score at Week 48 | 2.5 [-74 to 81] | 0.0 [-75 to 81]
Statistical Analysis 1: Comparison: DRV/Rtv 800/100 mg Once Daily vs DRV/Rtv 600/100 mg Twice Daily; Test type: Superiority or Other; p = 0.761, ANCOVA; Including factors for treatment, and baseline log10 plasma viral load and baseline FAHI score as covariates; Difference in least square means = 0.55, 95% CI 2-sided [-2.97 to 4.06], Standard Error of Mean 1.79 — Difference in least square means DRV/rtv once daily minus DRV/rtv twice daily estimated from the ANCOVA model

9. Secondary Outcome: Percentage of Participants Adherent/Non-adherent to ARV as Determined by Modified Medication Adherence Self Report Inventory (M-MASRI) Questionnaire at Week 48
Description: Self-reported adherence to the ARV medications was measured. The M-MASRI asks participants to report the number of doses taken, as well as the number of doses taken during the last 30 days prior to the study visit by means of a horizontal visual analogue scale (VAS) that generates a self-rated percentage of doses of all the ARV medications taken during the past 30 days.
Time Frame: 48 weeks
Population: Intent-to-Treat (ITT) population: Participants who were randomized and who received at least 1 dose of study medication.
Measure: Number; unit: Percentage of participants
Arm/Group | DRV/Rtv 800/100 mg Once Daily | DRV/Rtv 600/100 mg Twice Daily
Number analyzed (Participants) | 294 | 296
Percentage of participants
  Adherent | 67.4 | 60.3
  Non-adherent | 32.6 | 39.7

10. Secondary Outcome: Area Under the Curve From the Time of Study Medication Administration Upto 24 Hour Postdose (AUC24h) of DRV and Rtv
Description: Pharmacokinetic parameter AUC24h was assessed from the time of study medication administration upto 24 hour postdose. Population Pharmacokinetic Estimates of DRV and rtv were evaluated.
Time Frame: 0 hour predose and 1 hour post dose measured at Weeks 4 and 24. Any time point measured at Weeks 8 and 48.
Population: Intent-to-Treat (ITT) population: Participants who were randomized and who received at least 1 dose of study medication.
Measure: Median (Full Range); unit: ng*h/mL
Arm/Group | DRV/Rtv 800/100 mg Once Daily | DRV/Rtv 600/100 mg Twice Daily
Number analyzed (Participants) | 294 | 296
ng*h/mL
  Population Pharmacokinetic Estimates of DRV | 87788 [45456 to 236920] | 109401 [48934 to 323820]
  Population Pharmacokinetic Estimates of rtv | 5776 [1801 to 39027] | 12588 [3404 to 44762]

11. Secondary Outcome: Predose Plasma Concentration (C0h) of DRV and Rtv.
Description: Pharmacokinetic parameter C0h was assessed. Population Pharmacokinetic Estimates of DRV and rtv were evaluated.
Time Frame: 0 hour predose and 1 hour post dose measured at Weeks 4 and 24. Any time point measured at Weeks 8 and 48
Population: Intent-to-Treat (ITT) population: Participants who were randomized and who received at least 1 dose of study medication.
Measure: Median (Full Range); unit: ng/mL
Arm/Group | DRV/Rtv 800/100 mg Once Daily | DRV/Rtv 600/100 mg Twice Daily
Number analyzed (Participants) | 294 | 296
ng/mL
  Population Pharmacokinetic Estimates of DRV | 1896 [184 to 7881] | 3197 [250 to 11865]
  Population Pharmacokinetic Estimates of rtv | 59 [6 to 1049] | 307 [41 to 1657]

12. Secondary Outcome: Number of Participants Developing Mutations at Endpoint
Description: Development of Mutations in Virologic Failures (Plasma Viral Load less than 50 Copies/mL) at endpoint.
Time Frame: 48 weeks
Population: Intent-to-Treat (ITT) population: Participants who were randomized and who received at least 1 dose of study medication.
Measure: Number; unit: Participants
Arm/Group | DRV/Rtv 800/100 mg Once Daily | DRV/Rtv 600/100 mg Twice Daily
Number analyzed (Participants) | 294 | 296
Participants
  DRV resistance-associated mutation (RAM) | 1 | 0
  Primary (major) protease inhibitor (PI) mutations | 1 | 0
  Protease inhibitor (PI) RAMs | 7 | 4
  Nucleoside reverse transcriptase inhibitor RAMs | 4 | 3

ADVERSE EVENTS:
Time Frame: 52 weeks
Arm/Group | DRV/Rtv 800/100 mg Once Daily | DRV/Rtv 600/100 mg Twice Daily
Serious Adverse Events (participants affected / at risk) | 16/294 | 27/296
Other Adverse Events (participants affected / at risk) | 134/294 | 147/296
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | DRV/Rtv 800/100 mg Once Daily (N=294) | DRV/Rtv 600/100 mg Twice Daily (N=296)
Pneumonia (Infections and infestations) | 3 | 3
Dermo-hypodermitis (Infections and infestations) | 0 | 1
Escherichia urinary tract infection (Infections and infestations) | 0 | 1
Gastroenteritis cryptosporidial (Infections and infestations) | 0 | 1
Lung infection (Infections and infestations) | 0 | 1
Mastoiditis (Infections and infestations) | 0 | 1
Peritonitis bacterial (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 0 | 1
Toxoplasmosis (Infections and infestations) | 0 | 1
Appendicitis (Infections and infestations) | 1 | 0
Bronchopneumonia (Infections and infestations) | 1 | 0
Extrapulmonary tuberculosis (Infections and infestations) | 1 | 0
Infected cyst (Infections and infestations) | 1 | 0
Influenza (Infections and infestations) | 1 | 0
Lobar pneumonia (Infections and infestations) | 1 | 0
Malaria (Infections and infestations) | 1 | 0
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 | 1
Hyperamylasaemia (Metabolism and nutrition disorders) | 0 | 1
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 | 1
Lactic acidosis (Metabolism and nutrition disorders) | 0 | 1
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary bulla (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hypoventilation (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 2
Bicytopenia (Blood and lymphatic system disorders) | 0 | 1
Lymphadenopathy (Blood and lymphatic system disorders) | 1 | 0
Calculus ureteric (Renal and urinary disorders) | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 0 | 1
Renal failure acute (Renal and urinary disorders) | 0 | 1
Cardiac failure congestive (Cardiac disorders) | 0 | 2
Atrioventricular block first degree (Cardiac disorders) | 0 | 1
Sinus bradycardia (Cardiac disorders) | 0 | 1
Cardio-respiratory arrest (Cardiac disorders) | 1 | 0
Bile duct obstruction (Hepatobiliary disorders) | 0 | 1
Hepatitis (Hepatobiliary disorders) | 0 | 1
Alcohol poisoning (Injury, poisoning and procedural complications) | 0 | 1
Concussion (Injury, poisoning and procedural complications) | 0 | 1
Drug toxicity (Injury, poisoning and procedural complications) | 0 | 1
Skin laceration (Injury, poisoning and procedural complications) | 0 | 1
Whiplash injury (Injury, poisoning and procedural complications) | 0 | 1
Overdose (Injury, poisoning and procedural complications) | 1 | 0
Post procedural bile leak (Injury, poisoning and procedural complications) | 1 | 0
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Uterine cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Anxiety (Psychiatric disorders) | 0 | 2
Abnormal behaviour (Psychiatric disorders) | 0 | 1
Suicidal ideation (Psychiatric disorders) | 1 | 0
Suicide attempt (Psychiatric disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1
Drug interaction (General disorders) | 0 | 1
Pyrexia (General disorders) | 1 | 0
Weight decreased (Investigations) | 0 | 1
Carpal tunnel syndrome (Nervous system disorders) | 0 | 1
Carotid artery aneurysm (Nervous system disorders) | 1 | 0
Angiodermatitis (Skin and subcutaneous tissue disorders) | 0 | 1
Retinal detachment (Eye disorders) | 1 | 0
Vulval ulceration (Reproductive system and breast disorders) | 1 | 0
Intervertebral disc operation (Surgical and medical procedures) | 1 | 0
Deep vein thrombosis (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | DRV/Rtv 800/100 mg Once Daily (N=294) | DRV/Rtv 600/100 mg Twice Daily (N=296)
Diarrhoea (Gastrointestinal disorders) | 42 | 66
Nausea (Gastrointestinal disorders) | 38 | 42
Vomiting (Gastrointestinal disorders) | 13 | 25
Nasopharyngitis (Infections and infestations) | 19 | 19
Influenza (Infections and infestations) | 17 | 18
Upper respiratory tract infection (Infections and infestations) | 17 | 18
Bronchitis (Infections and infestations) | 16 | 11
Headache (Nervous system disorders) | 20 | 20
Rash (Skin and subcutaneous tissue disorders) | 15 | 14
Back pain (Musculoskeletal and connective tissue disorders) | 16 | 11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor will not unreasonably withhold consent to publish the data generated in this trial. However, it is the policy of the Sponsor not to allow the investigators to publish their results or findings prior to the Sponsor's publication of the overall trial results. The investigator agrees that before he/she publishes any results of this trial, he/she shall allow at least 45 days for the Sponsor to review the prepublication manuscript prior to submission of the manuscript to the publisher.